CLINICAL TRIAL: NCT00610896
Title: CRM and Fusion Beats: Effects of Progressive Fusion on Intra-left Ventricular Mechanical Function
Status: Completed | Type: Observational
Sponsor: Essentia Health (Other)
Responsible Party: Michael E. Mollerus, MD, Essentia Health
Other Study IDs: 12-07-02
Record Dates: First submitted 2008-01-25; First posted 2008-02-08 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: 30 Patients with dualchamber pacemakers or implantable cardioverter-defibrillators (ICDs)

SUMMARY:
This study is looking at cardiac rhythm management (CRM) and fusion beats in patients who have a pacemaker or implantable cardioverter-defibrillator (ICD), to determine if there is a correlation between the time between the contraction of the upper chambers of the heart (atrium) and the lower chambers of the heart, (ventricle) and heart function.

Some studies of people with pacemakers have been done to determine if shortening the time of contraction between the atrium and ventricle could benefit the function of the left ventricle. These studies have shown that there is no benefit in heart function.There have been other studies which have shown that chronic pacing of the right ventricle, especially with the lead placed at the tip of the right ventricle, can lead to a decrease in the function of the left ventricle and congestive heart failure. In some patients long term pacing of the right ventricle has also been associated with a reduction in the ability of the left ventricle to pump blood. This is know as a reduced left ventricular ejection fraction, which can be documented by an echocardiogram.

This study proposes to evaluate the acute effects of progressive paced fusion beats on the left ventricle to answer the question whether there is an delay between the atrium and ventricle that is "too long" or "too short".

ELIGIBILITY:
Inclusion Criteria:

* Dual chamber pacemaker or ICD device
* Left Ventrical Ejection Fraction (LVEF) 40% or less
* Sinus Rhythm with intact atrioventricular conduction with a PR interval greater than 200 msec QRS less than 120 msec
* Pacing right ventricle lead in the right ventricular apex (RVA), system implanted within 6 weeks or chronically implanted system with histograms showing 20% or less right ventricle pacing

Exclusion Criteria:

* LVEF greater than 40%,
* Any rhythm other than sinus rhythm
* Second degree or higher atrioventricular block
* Native Heart Rate less than 40 beats per minute or greater than 90 beats per minute
* Left ventricle or Chronic Sinus lead in non-RVA location
* Chronically implanted system with greater than 20% right ventricle pacing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pacemaker clinic or inpatient EP at St. Marys' Medical Center Duluth MN
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2008-01; Primary Completion 2010-05 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Acute effect of mechanical dyssynchrony measured by septal to lateral wall delay using tissue doppler imaging between baseline non-fused atrioventricular conduction and varying degrees of paced and native atrioventricular conduction.

SECONDARY OUTCOMES:
Stroke volume as measured by time velocity integral across the aorta valve between baseline non-fused atrioventricular conduction, and varying degrees of paced and native atrioventricular conduction.

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Mollerus, MD, Principal Investigator — Essentia Health
Locations (1):
- Essentia Health, Duluth, Minnesota, United States

REFERENCES:
- [Background] Auricchio A, Sommariva L, Salo RW, Scafuri A, Chiariello L. Improvement of cardiac function in patients with severe congestive heart failure and coronary artery disease by dual chamber pacing with shortened AV delay. Pacing Clin Electrophysiol. 1993 Oct;16(10):2034-43. doi: 10.1111/j.1540-8159.1993.tb00997.x. PMID 7694250
- [Background] Gold MR, Feliciano Z, Gottlieb SS, Fisher ML. Dual-chamber pacing with a short atrioventricular delay in congestive heart failure: a randomized study. J Am Coll Cardiol. 1995 Oct;26(4):967-73. doi: 10.1016/0735-1097(95)00292-0. PMID 7560625
- [Background] Shinbane JS, Chu E, DeMarco T, Sobol Y, Fitzpatrick AP, Lau DM, Klinski C, Schiller NB, Griffin JC, Chatterjee K. Evaluation of acute dual-chamber pacing with a range of atrioventricular delays on cardiac performance in refractory heart failure. J Am Coll Cardiol. 1997 Nov 1;30(5):1295-300. doi: 10.1016/s0735-1097(97)00307-0. PMID 9350930
- [Background] Sweeney MO, Hellkamp AS, Ellenbogen KA, Greenspon AJ, Freedman RA, Lee KL, Lamas GA; MOde Selection Trial Investigators. Adverse effect of ventricular pacing on heart failure and atrial fibrillation among patients with normal baseline QRS duration in a clinical trial of pacemaker therapy for sinus node dysfunction. Circulation. 2003 Jun 17;107(23):2932-7. doi: 10.1161/01.CIR.0000072769.17295.B1. Epub 2003 Jun 2. PMID 12782566
- [Background] Steinberg JS, Fischer A, Wang P, Schuger C, Daubert J, McNitt S, Andrews M, Brown M, Hall WJ, Zareba W, Moss AJ; MADIT II Investigators. The clinical implications of cumulative right ventricular pacing in the multicenter automatic defibrillator trial II. J Cardiovasc Electrophysiol. 2005 Apr;16(4):359-65. doi: 10.1046/j.1540-8167.2005.50038.x. PMID 15828875
- [Background] Thambo JB, Bordachar P, Garrigue S, Lafitte S, Sanders P, Reuter S, Girardot R, Crepin D, Reant P, Roudaut R, Jais P, Haissaguerre M, Clementy J, Jimenez M. Detrimental ventricular remodeling in patients with congenital complete heart block and chronic right ventricular apical pacing. Circulation. 2004 Dec 21;110(25):3766-72. doi: 10.1161/01.CIR.0000150336.86033.8D. Epub 2004 Dec 6. PMID 15583083
- [Background] Tse HF, Lau CP. Long-term effect of right ventricular pacing on myocardial perfusion and function. J Am Coll Cardiol. 1997 Mar 15;29(4):744-9. doi: 10.1016/s0735-1097(96)00586-4. PMID 9091519
- [Background] Lieberman R, Padeletti L, Schreuder J, Jackson K, Michelucci A, Colella A, Eastman W, Valsecchi S, Hettrick DA. Ventricular pacing lead location alters systemic hemodynamics and left ventricular function in patients with and without reduced ejection fraction. J Am Coll Cardiol. 2006 Oct 17;48(8):1634-41. doi: 10.1016/j.jacc.2006.04.099. Epub 2006 Sep 27. PMID 17045900
- [Background] Yu CM, Sanderson JE, Marwick TH, Oh JK. Tissue Doppler imaging a new prognosticator for cardiovascular diseases. J Am Coll Cardiol. 2007 May 15;49(19):1903-14. doi: 10.1016/j.jacc.2007.01.078. Epub 2007 Apr 30. PMID 17498573
- [Background] Bax JJ, Bleeker GB, Marwick TH, Molhoek SG, Boersma E, Steendijk P, van der Wall EE, Schalij MJ. Left ventricular dyssynchrony predicts response and prognosis after cardiac resynchronization therapy. J Am Coll Cardiol. 2004 Nov 2;44(9):1834-40. doi: 10.1016/j.jacc.2004.08.016. PMID 15519016
- [Background] Tops LF, Schalij MJ, Holman ER, van Erven L, van der Wall EE, Bax JJ. Right ventricular pacing can induce ventricular dyssynchrony in patients with atrial fibrillation after atrioventricular node ablation. J Am Coll Cardiol. 2006 Oct 17;48(8):1642-8. doi: 10.1016/j.jacc.2006.05.072. Epub 2006 Sep 27. PMID 17045901
- [Background] Catanzariti D, Maines M, Cemin C, Broso G, Marotta T, Vergara G. Permanent direct his bundle pacing does not induce ventricular dyssynchrony unlike conventional right ventricular apical pacing. An intrapatient acute comparison study. J Interv Card Electrophysiol. 2006 Aug;16(2):81-92. doi: 10.1007/s10840-006-9033-5. Epub 2006 Nov 18. PMID 17115267
- [Background] Victor F, Mabo P, Mansour H, Pavin D, Kabalu G, de Place C, Leclercq C, Daubert JC. A randomized comparison of permanent septal versus apical right ventricular pacing: short-term results. J Cardiovasc Electrophysiol. 2006 Mar;17(3):238-42. doi: 10.1111/j.1540-8167.2006.00358.x. PMID 16643392
- [Background] Stambler BS, Ellenbogen K, Zhang X, Porter TR, Xie F, Malik R, Small R, Burke M, Kaplan A, Nair L, Belz M, Fuenzalida C, Gold M, Love C, Sharma A, Silverman R, Sogade F, Van Natta B, Wilkoff BL; ROVA Investigators. Right ventricular outflow versus apical pacing in pacemaker patients with congestive heart failure and atrial fibrillation. J Cardiovasc Electrophysiol. 2003 Nov;14(11):1180-6. doi: 10.1046/j.1540-8167.2003.03216.x. PMID 14678131
- [Background] Olshansky B, Day JD, Moore S, Gering L, Rosenbaum M, McGuire M, Brown S, Lerew DR. Is dual-chamber programming inferior to single-chamber programming in an implantable cardioverter-defibrillator? Results of the INTRINSIC RV (Inhibition of Unnecessary RV Pacing With AVSH in ICDs) study. Circulation. 2007 Jan 2;115(1):9-16. doi: 10.1161/CIRCULATIONAHA.106.629428. Epub 2006 Dec 18. PMID 17179021
- [Background] Olshansky B, Day J, McGuire M, Hahn S, Brown S, Lerew DR. Reduction of right ventricular pacing in patients with dual-chamber ICDs. Pacing Clin Electrophysiol. 2006 Mar;29(3):237-43. doi: 10.1111/j.1540-8159.2006.00329.x. PMID 16606390
- [Background] Postaci N, Yesil M, Susam I, Bayata S. The influence of different AV delays on left ventricular diastolic functions and on incidence of diastolic mitral regurgitation. Angiology. 1996 Sep;47(9):895-9. doi: 10.1177/000331979604700908. PMID 8810656
- [Background] Jutzy RV, Feenstra L, Pai R, Florio J, Bansal R, Aybar R, Levine PA. Comparison of intrinsic versus paced ventricular function. Pacing Clin Electrophysiol. 1992 Nov;15(11 Pt 2):1919-22. doi: 10.1111/j.1540-8159.1992.tb02994.x. PMID 1279572
- [Background] Videen JS, Huang SK, Bazgan ID, Mechling E, Patton DD. Hemodynamic comparison of ventricular pacing, atrioventricular sequential pacing, and atrial synchronous ventricular pacing using radionuclide ventriculography. Am J Cardiol. 1986 Jun 1;57(15):1305-8. doi: 10.1016/0002-9149(86)90209-2. PMID 3717030
- [Background] Nielsen JC, Pedersen AK, Mortensen PT, Andersen HR. Programming a fixed long atrioventricular delay is not effective in preventing ventricular pacing in patients with sick sinus syndrome. Europace. 1999 Apr;1(2):113-20. doi: 10.1053/eupc.1998.0026. PMID 11228853
- [Background] de Cock CC, Giudici MC, Twisk JW. Comparison of the haemodynamic effects of right ventricular outflow-tract pacing with right ventricular apex pacing: a quantitative review. Europace. 2003 Jul;5(3):275-8. doi: 10.1016/s1099-5129(03)00031-x. PMID 12842643
- [Background] Wilkoff BL, Cook JR, Epstein AE, Greene HL, Hallstrom AP, Hsia H, Kutalek SP, Sharma A; Dual Chamber and VVI Implantable Defibrillator Trial Investigators. Dual-chamber pacing or ventricular backup pacing in patients with an implantable defibrillator: the Dual Chamber and VVI Implantable Defibrillator (DAVID) Trial. JAMA. 2002 Dec 25;288(24):3115-23. doi: 10.1001/jama.288.24.3115. PMID 12495391